CLINICAL TRIAL: NCT00525252
Title: Maintaining Alcohol Abstinence in Alcoholic Patients With Liver Cirrhosis: Efficacy and Safety of Baclofen Administration in a Randomized Double Blind Controlled Study
Brief Title: Efficacy of Baclofen in the Treatment of Alcohol Addiction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bacl001
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Liver Cirrhosis, Alcoholic
Keywords: Liver cirrhosis; Alcoholism; Craving
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Liver Cirrhosis; Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): A total of 42 alcoholic patients with liver cirrhosis treated with placebo
  Interventions: Drug: placebo
- 1 (Active Comparator): a total of 42 alcoholic patients with liver cirrhosis treated by baclofen
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Baclofen orally administered for 12 consecutive weeks. For the first 3 days, baclofen administered at a dose of 5 milligrams 3 times per day; subsequently, the daily dose of baclofen will be increased to 10 milligrams 3 times per day.
  Arms: 1
Drug: placebo — Placebo will be orally administered for 12 consecutive weeks
  Arms: 2

SUMMARY:
Intervention to achieve alcohol abstinence represents the most effective treatment for alcoholic patients with liver cirrhosis. However no trials have evaluated the efficacy of anti-craving drugs in these patients because of the concern that these medications might worsen liver disease. Baclofen is effective to reduce alcohol craving improving abstinence in alcohol-dependent patients. It is mainly eliminated by kidney. No hepatic side-effects have been reported in treated patients. The present study investigates the efficacy and safety of baclofen in achieving and maintaining abstinence in alcoholic cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18 to 75 years
* diagnosis of alcohol dependence according to DSM IV criteria
* diagnosis of liver cirrhosis
* alcohol intake of at least 2 heavy drinking days (men > 5 drinks/days; women > 4 drinks/day) per week, on average and an average overall consumption of 21 drinks/week or more for men and 14 drinks/week or more for women during the 4 weeks prior to enrolment
* presence of a referred family member

Exclusion Criteria:

* severe heart or lung disease
* kidney alterations and/or hepato-renal syndrome
* tumours, including hepatocellular carcinoma
* metabolic diseases, including diabetes
* clinical signs of hepatic encephalopathy
* patients treated with interferon or corticosteroids within the last 60 days
* psychopathological illness undergoing treatment with psychoactive drugs
* epilepsy or epileptiform convulsions
* addiction to drugs other than nicotine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2003-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Total alcohol abstinence; cumulative abstinence duration | 12 weeks

SECONDARY OUTCOMES:
Obsessive and Compulsive craving | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Addolorato, M.D., Principal Investigator — Catholic University of Rome

REFERENCES:
- [Background] Addolorato G, Caputo F, Capristo E, Domenicali M, Bernardi M, Janiri L, Agabio R, Colombo G, Gessa GL, Gasbarrini G. Baclofen efficacy in reducing alcohol craving and intake: a preliminary double-blind randomized controlled study. Alcohol Alcohol. 2002 Sep-Oct;37(5):504-8. doi: 10.1093/alcalc/37.5.504. PMID 12217947
- [Derived] Addolorato G, Leggio L, Ferrulli A, Cardone S, Vonghia L, Mirijello A, Abenavoli L, D'Angelo C, Caputo F, Zambon A, Haber PS, Gasbarrini G. Effectiveness and safety of baclofen for maintenance of alcohol abstinence in alcohol-dependent patients with liver cirrhosis: randomised, double-blind controlled study. Lancet. 2007 Dec 8;370(9603):1915-22. doi: 10.1016/S0140-6736(07)61814-5. PMID 18068515